CLINICAL TRIAL: NCT06089005
Title: Home-based Instrument-assisted Soft Tissue Mobilization for Pain Relief in Patients With Iliotibial Band Syndrome: A Prospective, Pre-post Intervention Study
Brief Title: Home-based Treatment Using the Sidekick Tool for Pain Relief in Patients With Iliotibial Band Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hannah Antony (Industry)
Responsible Party: Sponsor-Investigator, Hannah Antony, Product Education Lead, Sidekick In
Organization: Sidekick In (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIDEKICK101002
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Iliotibial Band Syndrome
Keywords: Iliotibial band friction syndrome; Iliotibial band pain
MeSH Terms: conditions — Iliotibial Band Syndrome

STUDY DESIGN:
Intervention Model Description: pre post test single group intervention study design
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): daily use of the IASTM on the hip, quad and glute muscles for 60s in duration each session
  Interventions: Device: Instrument Assisted Soft Tissue Mobilization device

INTERVENTIONS:
Device: Instrument Assisted Soft Tissue Mobilization device — Application of IASTM tool on specific muscle areas twice daily for intervention protocol of 7 days

SUMMARY:
The aim of the study is to test how well the Sidekick Tool works as a home-based pain relief for iliotibial band syndrome using instrument assisted soft tissue mobilization tool in healthy participants aged 18-65 years old. We hypothesize that the use of the tool over the course of seven days and by following a home-treatment plan will result in less pain that is caused by iliotibial band syndrome for the participants. Pain intensity will be measured using a Numerical Pain Rating Scale from 0-to-10. Other measurements will include pain intensity after exercise and if participants return to their sport.

Participants will be asked to complete an online questionnaire to ensure they are a good fit for the study. Once they have been entered into the study, they will complete a video call with the researchers to go gather their current pain intensity levels. Participants will be emailed the instructions for how to use the tool for seven days and will be mailed the Sidekick Tool to their home.

After seven days of using the tool, the participants will be asked to complete a final video call to gather their pain intensity levels. This number will be compared to their initial pain intensity to see if their pain has lowered while using the tool.

DETAILED DESCRIPTION:
The objective of the study is to provide evidence to support the home-based treatment of muscle scraping for iliotibial band syndrome (ITBS). The hypothesis of the researchers is that using the instrument assisted soft tissue mobilization (IASTM) tool provided by Sidekick, will result in reduced pain after following a home-treatment plan for seven days. The study aims to provide evidence for non-invasive treatments to reduce the healthcare costs and burden.

Prior to the commencement of the study, all the subjects selected signed an informed consent document, as defined by the Declaration of Helsinki. The sponsor is Sidekick Inc and the principal investigator is under direct employment of the sponsor.

The study is a single group, pre- post-test comparison, following STROBE guidelines on a group of 30-40 healthy participants. An incentive of $50 USD will be provided to the participants at completion of study, as well, the participants will get to keep the tool but are not told this.

The Sidekick tool used will be the Swerve, which will be mailed to participants once the eligibility questionnaire, informed consent, pre-test questionnaire and initial video call are completed. Participants will be informed to not start new pharmacological interventions, no new stretching, no in-person treatments with a clinician/healthcare professional during the seven day intervention period. Participants will use a tracker to monitor use of the tool and pain responses.

Participants will receive the following detailed instructions for use of the Sidekick tool:

For all locations, use a moderate but comfortable pressure. Frequency: two sessions daily, morning and night. Duration: 3 minutes total duration in each session.

Steps to complete muscle scraping on the tensor fascia latae, vastus lateralis and glute muscles will all state the following steps: Set a timer ready for 60s. Rub the pump gel on the muscle, or complete muscle scraping over tight clothing. You will use the Swerve tool on the stated muscle.

Fill in the Sidekick Tracker to monitor your use of the tool, what time of day and sensations felt during and after completing the protocol A reminder for safety considerations including repeating contraindications, and instructions on what to do if adverse events such as petechiae or ecchymosis occur during using the tool: Pressure should be firm but comfortable, it may produce skin redness but shouldn't produce a blanket red color, if so, reduce pressure or end the session on that muscle group If post-treatment bruising occurs, stop the intervention until it completely heals and the skin returns to it's pre-treatment color.

A mid way follow up and check in via email will be conducted to ensure participants are following the protocol and to take note of any adverse reactions. After seven days, a final video call will be conducted and the participants will fill out the post-test questionnaire.

Within-group changes from baseline will be tested with paired Student's t-tests. Two-sided P-values < 0.05 were considered statistically significant. All analyses will be performed in R (version 4.1.2, Vienna, Austria).

ELIGIBILITY:
Inclusion Criteria:

* diagnosed (have them enter the month of diagnosis) by a physician or physical therapist
* pain on lateral side of knee
* tenderness on palpation at lateral knee
* unilateral symptoms only
* past treatments can include rolling, stretching
* pain duration of 3-12 weeks

Exclusion Criteria:

* bilateral symptoms
* no diagnosis
* other knee pain conditions
* prior surgeries of the lower limb
* current pharmacological treatments

Any contraindications including:

open wounds or unhealed sites Thrombophlebitis uncontrolled hypertension or high blood pressure skin infections Current hematoma myositis ossificans Boney fractures high pain sensation acute inflammatory conditions congestive heart disease circulatory disorders Osteoporosis Cancer Pregnancy Type 1 diabetes Type 2 diabetes varicose veins kidney dysfunction rheumatoid arthritis Lymphedema chronic regional pain syndrome Current use of steroidal medications Current use of anticoagulant medications Current use of NSAID medications (non-steroidal anti-inflammatory drugs)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-23 (Estimated); Primary Completion 2023-11-24 (Estimated); Study Completion 2023-11-24 (Estimated)

PRIMARY OUTCOMES:
Pain intensity during the day | Day 0, Day 7
  Numerical pain rating scale 0-to-10

SECONDARY OUTCOMES:
Pain intensity after exercise | Day 0, Day 7
  Numerical pain rating scale 0-to-10
Return to sport | Day 0, day 7
  Yes, no binary option participant count
Number of participants with adverse effects after use of intervention | Day 0, Day 7
  Yes, no binary option participant count